CLINICAL TRIAL: NCT03583385
Title: A Randomized, Open-label, Two-way Crossover Study Assessing the Bioequivalence (BE) Between Single Dose of 750 mg Glucophage® XR Tablets (PT Merck Tbk, Jakarta, Indonesia-Manufactured) and 750 mg Glucophage® XR Tablets (Merck Santé, Semoy, France-Manufactured) Under Fasted State in Healthy Subjects
Brief Title: Glucophage® Extended Release (XR) 750 Milligram (mg) Indonesia Bioequivalence (BE) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: MS200084_0015
Record Dates: First submitted 2018-06-28; First posted 2018-07-11 (Actual); Results first posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin; Drug Evaluation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Glucophage XR (Test), Then Glucophage XR (Comparator) (Experimental): Participants received single oral dose of 750 milligram (mg) Glucophage® XR tablet manufactured by PT Merck Tbk, Jakarta, Indonesia (Test Drug) in treatment period 1 followed by single oral dose of 750 mg Glucophage® XR tablet manufactured by Merck Santé, Semoy, France (Comparator Drug) in treatment period 2 under fasting conditions. The two periods were separated by a 7-day wash-out period.
  Interventions: Drug: Glucophage XR (Test drug); Drug: Glucophage XR (Comparator drug)
- First Glucophage XR (Comparator), Then Glucophage XR (Test) (Experimental): Participants received single oral dose of 750 milligram (mg) Glucophage® XR tablet manufactured by Merck Santé, Semoy, France (Comparator Drug) in treatment period 1 followed by single oral dose of 750 mg Glucophage® XR tablet manufactured by PT Merck Tbk, Jakarta, Indonesia (Test Drug) in treatment period 2 under fasting conditions. The two periods were separated by a 7-day wash-out period.
  Interventions: Drug: Glucophage XR (Test drug); Drug: Glucophage XR (Comparator drug)

INTERVENTIONS:
Drug: Glucophage XR (Test drug) — Participants received single oral dose of Glucophage® XR tablet manufactured by PT Merck Tbk, Jakarta, Indonesia (Test Drug) under fasted conditions.
  Other Names: Metformin hydrochloride
Drug: Glucophage XR (Comparator drug) — Participants received single oral dose of Glucophage® XR tablet manufactured by Merck Santé, Semoy, France (Comparator Drug) under fasted conditions.
  Other Names: Metformin hydrochloride

SUMMARY:
The purpose of this study is to assess bioequivalence between metformin hydrochloride (Glucophage® XR) manufactured in PT Merck Tbk, Indonesia (test drug) and metformin hydrochloride (Glucophage® XR) manufactured in Merck Santé, France (comparator drug) following single oral dose administration under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Participants has provided written informed consent prior to the conduct of any study-related activities
* Body mass index of 18 to 25 kilogram per square meter (kg/m^2)
* Good physical and mental health status, determined on the basis of medical history and physical examination
* Vital signs (blood pressure, pulse rate, respiratory rate and body temperature) in sitting position within the normal range or showing no clinically relevant deviation per the Investigator's opinion
* All values for laboratory assessments (hematology, clinical chemistry and urinalysis) within the normal range or showing no clinically relevant deviation per the Investigator's opinion
* No clinically significant abnormality on 12-lead electrocardiogram (ECG) recording as judged by the Investigator; corrected QT interval (QTc) (Bazett) should be less than equals to (<=) 450 milliseconds (ms)
* Non-smoker or smoker less than 10 cigarettes per day
* Women of childbearing potential (WOCBP) who are not nursing, are not pregnant, and are using highly effective methods of birth control. Female participants may also be enrolled if they are postmenopausal or surgically sterilized/ hysterectomized at least 6 months prior to study participation
* WOCBP must have a negative urine pregnancy test at Screening and on each admission (Day 1 of each dosing period)
* Negative screen for alcohol and drugs abuse (opiate class, barbiturates, cocaine and metabolites, amphetamines, cannabinoids and benzodiazepines) at Screening and on each Study Check-In (Day -1 of each dosing period)
* Negative screen for Hepatitis B surface antigen (HBsAg), Hepatitis C Virus (HCV) antibodies and/or Human Immunodeficiency Virus (HIV) antibodies.

Exclusion Criteria:

* Participation in a clinical trial/study within 90 days prior to Screening
* Blood donation (equal or more than 300 milliliter [mL]) or significant blood loss within 90 days prior to first drug administration
* Any surgical or medical condition, including findings in the medical history or in the prestudy assessments, or any other significant disease, that in the opinion of the investigator, constitutes a risk or a contraindication for the participation of the participant in the study or that could interfere with the study objectives, conduct or evaluation
* History of malignant diseases, except in-situ basal cell skin tumors treated with curative intent
* History of surgery of the gastrointestinal tract which could influence the gastrointestinal absorption and/or motility per the Investigator's opinion
* History or presence of relevant liver diseases or hepatic dysfunction (laboratory result for liver function test greater than equals to (>=) 1.5 upper limit of normal (ULN)
* History or presence of renal failure or renal dysfunction based on clinical symptoms and finding (serum creatinine concentration >1.4 milligram per milliliter (mg/mL)
* Ascertained or presumptive hypersensitivity to the active drug substance and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
* Receipt of any prescription or non-prescription medication within 14 days before the first drug administration, except for hormonal contraceptives in female, and including multivitamins and herbal products (e.g. St John's Wort)
* Consumption of large quantities of methylxanthine-containing beverages (> 5 cups of coffee/day or equivalent)
* Consumption of grapefruit, orange, cranberry or juices of these three fruits, 24 hours prior to drug administration
* Known lack of participant compliance or inability to communicate or cooperate with the Investigator (e.g., language problem, poor mental status)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — PT Merck Tbk, Indonesia, and affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- PT Equilab International, Jakarta, Indonesia

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | First Glucophage XR (Test), Then Glucophage XR (Comparator) | First Glucophage XR (Comparator), Then Glucophage XR (Test)
Started | 24 | 24
Completed | 23 | 23
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Treatment Period 2
Arm/Group | First Glucophage XR (Test), Then Glucophage XR (Comparator) | First Glucophage XR (Comparator), Then Glucophage XR (Test)
Started | 22 (Of 46 participants who completed period 1, 45 entered period2 & 1 participant didn't attend period2.) | 23
Completed | 21 | 23
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received Glucophage® XR 750 mg Tablet manufactured by PT Merck Tbk, Jakarta, Indonesia or Glucophage® XR 750 mg Tablet manufactured by Merck Santé, Semoy, France on Day 1 in either first treatment period or second treatment period.
Arm/Group | All Participants
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 48
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metformin
Description: The maximum plasma concentration of Metformin.
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: Pharmacokinetic (PK) analysis set included all participants without any relevant protocol deviations with respect to PK and absence of factors likely to affect the comparability of PK results, with adequate study medication compliance, and who have valid primary endpoints for both treatment.
Measure: Mean (Standard Deviation); unit: Nano-gram per milliliter (ng/mL)
Groups:
- Glucophage XR (Test): All participants who received Glucophage® XR 750 mg Tablet manufactured by PT Merck Tbk, Jakarta, Indonesia on Day 1 in either first treatment period or second treatment period.
- Glucophage XR (Comparator): All participants who received Glucophage® XR 750 mg Tablet (manufactured by Merck Santé, Semoy, France) on Day 1 in either first treatment period or second treatment period.
Arm/Group | Glucophage XR (Test) | Glucophage XR (Comparator)
Number analyzed (Participants) | 43 | 43
Nano-gram per milliliter (ng/mL) | 1109 (318.4) | 1087 (336.3)
Statistical Analysis 1: Comparison: Glucophage XR (Test) vs Glucophage XR (Comparator); Test type: Equivalence — Bio-equivalence Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.00% - 125.00%; % Ratio of Geometric Means = 103.42, 90% CI 2-sided [95.18 to 112.37]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Metformin
Description: Area under the plasma concentration-time curve from zero to the time of the last quantifiable concentration.
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: PK analysis set included all participants without any relevant protocol deviations with respect to PK and absence of factors likely to affect the comparability of PK results, with adequate study medication compliance, and who have valid primary endpoints for both treatment.
Measure: Mean (Standard Deviation); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Glucophage XR (Test) | Glucophage XR (Comparator)
Number analyzed (Participants) | 43 | 43
Nanogram*hour per milliliter (ng*h/mL) | 7387 (2535.7) | 6977 (2512.0)
Statistical Analysis 1: Comparison: Glucophage XR (Test) vs Glucophage XR (Comparator); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; % Ratio of Geometric Means = 106.78, 90% CI 2-sided [98.99 to 115.19]

3. Secondary Outcome: Area Under Plasma Concentration Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Metformin
Description: AUC (0-inf) is defined as the area under the plasma concentration versus time curve (AUC) from time zero (predose) to extrapolated infinite time (0-inf).
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Glucophage XR (Test) | Glucophage XR (Comparator)
Number analyzed (Participants) | 43 | 43
ng*h/mL | 7678 (2559.5) | 7250 (2523.6)

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Metformin
Description: Time of the maximum drug concentration.
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Glucophage XR (Test) | Glucophage XR (Comparator)
Number analyzed (Participants) | 43 | 43
Hours | 3.50 [2.00 to 6.00] | 3.00 [1.50 to 6.00]

5. Secondary Outcome: Terminal Elimination Half-life in Plasma (t½) of Metformin
Description: Elimination Half Life (t1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half.
Time Frame: Pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 7, 8, 10, 12, 16, 24, and 32 hours post-dose on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Glucophage XR (Test) | Glucophage XR (Comparator)
Number analyzed (Participants) | 43 | 43
Hours | 5.82 (2.875) | 6.03 (3.292)

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. Number of participants with TEAEs included participants with both non serious and serious TEAEs.
Time Frame: Up to Day 51
Population: The safety analysis set included all participants who have received at least one dose of the investigational product and have had one subsequent safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Glucophage XR (Test) | Glucophage XR (Comparator)
Number analyzed (Participants) | 47 | 46
Participants
  Treatment Emergent Adverse Events (TEAEs) | 5 | 9
  Serious TEAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 51
Description: The safety analysis set included all participants who have received at least one dose of the investigational product and have had one subsequent safety assessment.
Arm/Group | Glucophage XR (Test) | Glucophage XR (Comparator)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46
Other Adverse Events (participants affected / at risk) | 5/47 | 9/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glucophage XR (Test) (N=47) | Glucophage XR (Comparator) (N=46)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Stools loose (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 4
Headache (Nervous system disorders) | 4 | 7
Vomiting (Gastrointestinal disorders) | 0 | 1
Dermatitis venenata (Skin and subcutaneous tissue disorders) | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1
Urinary tract bleed microscopic (Renal and urinary disorders) | 1 | 1
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT03583385/SAP_000.pdf
  • Study Protocol (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT03583385/Prot_001.pdf